CLINICAL TRIAL: NCT01277523
Title: A Randomised, Double-blind, Placebo-controlled, Parallel-group Trial to Evaluate Efficacy and Safety of Tiotropium Inhalation Solution Delivered Via Respimat® Inhaler (2.5 mcg and 5 mcg Once Daily) Over 12 Weeks as add-on Controller Therapy on Top of Usual Care in Adolescents (12 to 17 Years Old) With Severe Persistent Asthma
Brief Title: Efficacy and Safety of 2 Doses of Tiotropium Respimat Compared to Placebo in Adolescents With Severe Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.456; 2010-021778-13 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide

ARMS (3):
- A (Experimental)
  Interventions: Drug: tiotropium low dose
- B (Experimental)
  Interventions: Drug: tiotropium high dose
- C (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tiotropium high dose — 2 actuations once daily
  Arms: B
Drug: placebo — 2 actuations once daily
  Arms: C
Drug: tiotropium low dose — 2 actuations once daily
  Arms: A

SUMMARY:
The overall purpose of the trial is to evaluate efficacy and safety of tiotropium inhalation solution delivered via Respimat® inhaler (2.5 mcg and 5 mcg once daily) over 12 weeks, compared to placebo, as add-on controller therapy on top of usual care in adolescents (12 to 17 years old) with severe persistent asthma.

The primary objective of the trial is to demonstrate superiority of tiotropium (5 mcg and possibly 2.5 mcg once daily in the evening) over placebo with regard to the primary pulmonary function endpoint after 12 weeks of treatment.

Secondary objectives are to evaluate efficacy of tiotropium with regard to other endpoints, and to evaluate the safety of tiotropium, compared to placebo, as add-on controller therapy on top of usual care in this patient population.

ELIGIBILITY:
Inclusion criteria:

1. All patients and their parent(s) (or legally accepted representative) must sign and date respectively an informed assent and an informed consent consistent with International Conference on Harmonisation - Harmonised Tripartite Guideline for Good Clinical Practice (ICH-GCP) guidelines and local legislation prior to the patient's participation in the trial. A separate informed consent/assent is required for pharmacogenomic sampling.
2. Male or female patients between 12 and 17 years of age (at date of informed consent/assent).
3. All patients must have at least a 3-month history of asthma at the time of enrolment into the trial.
4. All patients must have been on maintenance treatment with an inhaled corticosteroid either at stable high dose in combination with another controller medication, OR at stable medium dose in combination with two other controller medications, for at least 4 weeks before Visit 1.
5. All patients must be symptomatic at Visit 1 (screening) and prior to randomisation at Visit 2 as defined by an Asthma Control Questionnaire (ACQ) mean score of = 1.5.
6. All patients must have a pre-bronchodilator Forced Expiratory Volume in 1 second (FEV1) = 60% and = 90% of predicted normal at Visit 1.
7. Variation of absolute FEV1 values of Visit 1 (pre-bronchodilator, considered as 100%) as compared to Visit 2 (pre-dose) must be within ± 30%.
8. All patients must confirm the diagnosis of asthma by bronchodilator reversibility at Visit 1, resulting in an increase in FEV1 of = 12% and = 200 mL 15 to 30 minutes after 400 µg salbutamol (albuterol). If patients in the lower age range (e.g. 12 to 14 year old patients) exhibit a very small total lung volume, positive reversibility testing might be based solely on the relative (=12%) post-bronchodilator response.
9. All patients must be never-smokers or ex-smokers who stopped smoking at least one year prior to enrolment.
10. Patients must be able to use the Respimat® inhaler correctly.
11. Patients must be able to perform all trial related procedures including technically acceptable spirometric manoeuvres according to American Thoracic Society/ European Respiratory Society (ATS/ERS) standards and use of the electronic diary/peak flow meter (diary compliance of at least 80% is required).

Exclusion criteria:

1. Significant disease other than asthma.
2. Abnormal haematology or blood chemistry.
3. History of heart disease, and/or hospitalised for cardiac syncope or failure.
4. Any unstable or life-threatening or requiring intervention or cardiac arrhythmia.
5. Malignancy for which the patient has undergone resection, radiation therapy or chemotherapy.
6. Active tuberculosis.
7. Alcohol or drug abuse.
8. Thoracotomy with pulmonary resection.
9. Pulmonary rehabilitation program.
10. Hypersensitivity to anticholinergic drugs, or any components of the study medication delivery system.
11. Pregnant or nursing adolescent female patients.
12. Female patients of child-bearing potential not using a highly effective method of birth control.
13. Investigational drug within four weeks or six half lives prior to Visit 1.
14. Long-acting anticholinergics within four weeks prior to Visit 1.
15. Systemic corticosteroids at a high dose or at a not stable low dose within four weeks prior to Visit 1.
16. Leukotriene modifiers if not stabilised for at least four weeks prior to Visit 1.
17. Long-acting theophylline preparations if not stabilised for at least two weeks prior to Visit 1.
18. Anti Immunoglobulin E (Anti-IgE) treatment if not stabilised for at least six months prior to Visit 1.
19. Cromones if not stabilised within four weeks prior to Visit 1.
20. Oral beta-blocker medication within four weeks prior to Visit 1.
21. Systemic oral or i.v. or s.c. beta-adrenergics within four weeks prior to Visit 1.
22. Other non-approved and according to international guidelines not recommended experimental drugs for routine asthma therapy within four weeks prior to Visit 1.
23. Any acute asthma exacerbation or respiratory tract infection in the four weeks prior to Visit 1and/or in the four weeks prior to Visit 2. In case of an asthma deterioration occurring in the four weeks prior to Visit 1 and/or in the four weeks prior to Visit 2, the visit must be postponed.
24. Randomised in this trial or currently participating in another trial.
25. Narrow-angle glaucoma, or any other disease where anticholinergic treatment is contraindicated.
26. Moderate to severe renal impairment.
27. Patients requiring 10 or more puffs of rescue medication per day on more than 2 consecutive days in the four weeks prior to Visit 1 and/or in the four weeks prior to Visit 2. In case of an asthma deterioration occurring in the four weeks prior to Visit 1 and/or in the four weeks prior to Visit 2, the visit must be postponed.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 392 (Actual)
Dates: Start 2011-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (69):
- United States (8):
  - 205.456.01004 Boehringer Ingelheim Investigational Site, Stockton, California
  - 205.456.01008 Boehringer Ingelheim Investigational Site, Normal, Illinois
  - 205.456.01003 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 205.456.01007 Boehringer Ingelheim Investigational Site, Columbia, Missouri
  - 205.456.01002 Boehringer Ingelheim Investigational Site, Bellevue, Nebraska
  - 205.456.01001 Boehringer Ingelheim Investigational Site, Rockville Centre, New York
  - 205.456.01005 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 205.456.01006 Boehringer Ingelheim Investigational Site, Summerville, South Carolina
- Argentina (7):
  - 205.456.54002 Boehringer Ingelheim Investigational Site, Capital Federal
  - 205.456.54006 Boehringer Ingelheim Investigational Site, Capital Federal
  - 205.456.54008 Boehringer Ingelheim Investigational Site, Capital Federal
  - 205.456.54005 Boehringer Ingelheim Investigational Site, Mendoza
  - 205.456.54003 Boehringer Ingelheim Investigational Site, San Juan Bautista
  - 205.456.54004 Boehringer Ingelheim Investigational Site, San Miguel de Tucumán
  - 205.456.54009 Boehringer Ingelheim Investigational Site, San Miguel de Tucumán
- Australia (2):
  - 205.456.61002 Boehringer Ingelheim Investigational Site, Parkville, Victoria
  - 205.456.61001 Boehringer Ingelheim Investigational Site, Perth, Western Australia
- Bulgaria (3):
  - 205.456.35902 Boehringer Ingelheim Investigational Site, Plovdiv
  - 205.456.35901 Boehringer Ingelheim Investigational Site, Rousse
  - 205.456.35903 Boehringer Ingelheim Investigational Site, Sofia
- Germany (8):
  - 205.456.49008 Boehringer Ingelheim Investigational Site, Berlin
  - 205.456.49001 Boehringer Ingelheim Investigational Site, Bochum
  - 205.456.49004 Boehringer Ingelheim Investigational Site, Frankfurt
  - 205.456.49005 Boehringer Ingelheim Investigational Site, Kehl
  - 205.456.49003 Boehringer Ingelheim Investigational Site, Koblenz
  - 205.456.49010 Boehringer Ingelheim Investigational Site, Mainz
  - 205.456.49007 Boehringer Ingelheim Investigational Site, Neu-Isenburg
  - 205.456.49002 Boehringer Ingelheim Investigational Site, Wesel
- Guatemala (4):
  - 205.456.50201 Boehringer Ingelheim Investigational Site, Guatemala City
  - 205.456.50203 Boehringer Ingelheim Investigational Site, Guatemala City
  - 205.456.50204 Boehringer Ingelheim Investigational Site, Guatemala City
  - 205.456.50205 Boehringer Ingelheim Investigational Site, Guatemala City
- Hungary (6):
  - 205.456.36005 Boehringer Ingelheim Investigational Site, Budapest
  - 205.456.36002 Boehringer Ingelheim Investigational Site, Debrecen
  - 205.456.36004 Boehringer Ingelheim Investigational Site, Gyula
  - 205.456.36001 Boehringer Ingelheim Investigational Site, Miskolc
  - 205.456.36007 Boehringer Ingelheim Investigational Site, Mosdós
  - 205.456.36006 Boehringer Ingelheim Investigational Site, Nagyatád
- Israel (3):
  - 205.456.97205 Boehringer Ingelheim Investigational Site, Holon
  - 205.456.97203 Boehringer Ingelheim Investigational Site, Petah Tikva
  - 205.456.97201 Boehringer Ingelheim Investigational Site, Safed
- Latvia (5):
  - 205.456.37101 Boehringer Ingelheim Investigational Site, Baldone
  - 205.456.37104 Boehringer Ingelheim Investigational Site, Balvi
  - 205.456.37103 Boehringer Ingelheim Investigational Site, Rēzekne
  - 205.456.37102 Boehringer Ingelheim Investigational Site, Riga
  - 205.456.37105 Boehringer Ingelheim Investigational Site, Talsi
- Mexico (4):
  - 205.456.52001 Boehringer Ingelheim Investigational Site, Hermosillo Sonora
  - 205.456.52002 Boehringer Ingelheim Investigational Site, Monterrey
  - 205.456.52003 Boehringer Ingelheim Investigational Site, Monterrey
  - 205.456.52004 Boehringer Ingelheim Investigational Site, Nuevo León
- Philippines (2):
  - 205.456.09001 Boehringer Ingelheim Investigational Site, Quezon City
  - 205.456.09002 Boehringer Ingelheim Investigational Site, Quezon City
- Portugal (5):
  - 205.456.35105 Boehringer Ingelheim Investigational Site, Coimbra
  - 205.456.35101 Boehringer Ingelheim Investigational Site, Lisbon
  - 205.456.35102 Boehringer Ingelheim Investigational Site, Lisbon
  - 205.456.35104 Boehringer Ingelheim Investigational Site, Lisbon
  - 205.456.35103 Boehringer Ingelheim Investigational Site, Porto
- South Africa (2):
  - 205.456.27001 Boehringer Ingelheim Investigational Site, Cape Town
  - 205.456.27002 Boehringer Ingelheim Investigational Site, Durban
- Ukraine (10):
  - 205.456.38006 Boehringer Ingelheim Investigational Site, Dnipropetrovsk
  - 205.456.38004 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.456.38003 Boehringer Ingelheim Investigational Site, Kiev
  - 205.456.38010 Boehringer Ingelheim Investigational Site, Kryvyi Rih
  - 205.456.38009 Boehringer Ingelheim Investigational Site, Kyiv
  - 205.456.38001 Boehringer Ingelheim Investigational Site, Lviv
  - 205.456.38007 Boehringer Ingelheim Investigational Site, Lviv
  - 205.456.38005 Boehringer Ingelheim Investigational Site, Uzhhorod
  - 205.456.38008 Boehringer Ingelheim Investigational Site, Vinnytsia
  - 205.456.38002 Boehringer Ingelheim Investigational Site, Zaporizhzhya

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Halpin DMG, Meltzer EO, Pisternick-Ruf W, Moroni-Zentgraf P, Engel M, Zaremba-Pechmann L, Casale T, FitzGerald JM. Peak expiratory flow as an endpoint for clinical trials in asthma: a comparison with FEV1. Respir Res. 2019 Jul 18;20(1):159. doi: 10.1186/s12931-019-1119-6. PMID 31319851
- [Derived] Hamelmann E, Bernstein JA, Vandewalker M, Moroni-Zentgraf P, Verri D, Unseld A, Engel M, Boner AL. A randomised controlled trial of tiotropium in adolescents with severe symptomatic asthma. Eur Respir J. 2017 Jan 11;49(1):1601100. doi: 10.1183/13993003.01100-2016. Print 2017 Jan. PMID 27811070

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Respimat: Inhalation of placebo solution once daily for 12 weeks delivered by the Respimat Inhaler, as add on therapy on top of usual care.
- Tio R2.5: Inhalation of 2.5mcg tiotropium bromide solution once daily for 12 weeks delivered by the Respimat Inhaler, as add on therapy on top of usual care.
- Tio R5: Inhalation of 5mcg tiotropium bromide solution once daily for 12 weeks delivered by the Respimat Inhaler, as add on therapy on top of usual care.
Period: Overall Study
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Started | 135 | 127 | 130
Completed | 132 | 126 | 130
Not Completed | 3 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Other Reason not Defined | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set which included all randomised patients who were dispensed and received, at least one documented dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5 | Total
Number analyzed (Participants) | 135 | 127 | 130 | 392
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (1.7) | 14.4 (1.8) | 14.3 (1.6) | 14.2 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 47 | 47 | 150
  Male | 79 | 80 | 83 | 242

OUTCOME MEASURES:

1. Primary Outcome: FEV1 peak0-3 Change From Baseline
Description: Change from baseline in peak forced expiratory volume in 1 second within the first 3 hours post dosing (FEV1 peak0-3) measured at week 12.
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: Full Analysis Set (FAS) was the same as the treated set which included all randomised patients who were dispensed and received at least one documented dose of trial medication. Missing data at a visit was imputed by the available data from the patient at that visit. Completely missing data were handled by the statistical model.
Measure: Mean (Standard Error); unit: litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 132 | 126 | 130
litres | 0.438 (0.045) | 0.550 (0.046) | 0.528 (0.045)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.0457, Mixed Models Analysis — Stepwise testing of the null hypothesis was used to test the efficacy of Tio R5 and then Tio R2.5, each over placebo; Mean Difference (Final Values) = 0.111, 95% CI 2-sided [0.002 to 0.220], Standard Error of Mean 0.055 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.1039, Mixed Models Analysis — Stepwise testing of the null hypothesis was used to test the efficacy of Tio R5 and then Tio R2.5, each over placebo; Mean Difference (Final Values) = 0.090, 95% CI 2-sided [-0.019 to 0.198], Standard Error of Mean 0.055 — Difference calculated as Tio R5 minus placebo

2. Secondary Outcome: Trough FEV1 Change From Baseline
Description: Change from baseline in Trough (pre-dose) Forced expiratory volume in 1 second (FEV1) measured at week 12.
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 132 | 126 | 130
litres | 0.230 (0.048) | 0.345 (0.048) | 0.284 (0.048)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.0509, Mixed Models Analysis — Stepwise testing of the null hypothesis was used to test the efficacy of Tio R5 and then Tio R2.5, each over placebo; Mean Difference (Final Values) = 0.115, 95% CI 2-sided [-0.000 to 0.231], Standard Error of Mean 0.059 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.3605, Mixed Models Analysis — Stepwise testing of the null hypothesis was used to test the efficacy of Tio R5 and then Tio R2.5, each over placebo; Mean Difference (Final Values) = 0.054, 95% CI 2-sided [-0.061 to 0.168], Standard Error of Mean 0.058 — Difference calculated as Tio R5 minus placebo

3. Secondary Outcome: FVC peak0-3 Change From Baseline
Description: Change from baseline in Maximum forced vital capacity (FVC) measured within the first 3 hours after administration of trial medication (FVC peak0-3h) after 12 weeks of treatment.
  The measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 132 | 126 | 130
Litres | 0.279 (0.048) | 0.370 (0.049) | 0.342 (0.048)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.1264, Mixed Models Analysis; Mean Difference (Final Values) = 0.091, 95% CI 2-sided [-0.026 to 0.207], Standard Error of Mean 0.059 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.2845, Mixed Models Analysis; Mean Difference (Final Values) = 0.063, 95% CI 2-sided [-0.053 to 0.179], Standard Error of Mean 0.059 — Difference calculated as Tio R5 minus placebo

4. Secondary Outcome: FEV1 AUC (0-3h) Change From Baseline
Description: Change from baseline of area under the curve (AUC) from 0 to 3 hours for FEV1 (FEV1 AUC 0-3h) after 12 weeks of treatment. The AUC was calculated by using the trapezoidal rule divided by the observation time (3h).
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 10 mins before drug administration and 30 mins, 1 hour (h), 2h, 3h after drug administration at 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 132 | 126 | 130
Litres | 0.336 (0.043) | 0.449 (0.043) | 0.423 (0.043)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.0338, Mixed Models Analysis; Mean Difference (Final Values) = 0.113, 95% CI 2-sided [0.009 to 0.217], Standard Error of Mean 0.053 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.0999, Mixed Models Analysis; Mean Difference (Final Values) = 0.087, 95% CI 2-sided [-0.017 to 0.191], Standard Error of Mean 0.053 — Difference calculated as Tio R5 minus placebo

5. Secondary Outcome: FVC AUC (0-3h) Change From Baseline
Description: Change from baseline of area under the curve (AUC) from 0 to 3 hours for FVC (Forced vital capacity) (FVC AUC0-3h) after 12 weeks of treatment. The AUC was calculated by using the trapezoidal rule divided by the observation time (3h).
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 10 mins before drug administration and 30 mins, 1 hour (h), 2h, 3h after drug administration at 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 132 | 126 | 130
litres | 0.175 (0.045) | 0.262 (0.047) | 0.227 (0.046)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.1252, Mixed Models Analysis; Mean Difference (Final Values) = 0.087, 95% CI 2-sided [-0.024 to 0.198], Standard Error of Mean 0.057 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.3549, Mixed Models Analysis; Mean Difference (Final Values) = 0.052, 95% CI 2-sided [-0.058 to 0.163], Standard Error of Mean 0.056 — Difference calculated as Tio R5 minus placebo

6. Secondary Outcome: Control of Asthma as Assessed by ACQ6 Score.
Description: Change from baseline in Asthma Control Questionnaire (ACQ) 6 score measured at week 12
  The ACQ is a scale containing 7 questions, each question has a 7 point scale which ranges from 0 to 6. A score of 0 corresponds to no impairment and a score of 6 corresponds to maximum impairment. ACQ6 score is calculated as the mean of the responses to the first 6 questions of the ACQ6.
  The measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 132 | 126 | 130
units on a scale | 1.144 (0.069) | 1.262 (0.071) | 1.197 (0.070)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.1819, Mixed Models Analysis; Mean Difference (Final Values) = 0.118, 95% CI 2-sided [-0.055 to 0.292], Standard Error of Mean 0.088 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.5448, Mixed Models Analysis; Mean Difference (Final Values) = 0.053, 95% CI 2-sided [-0.119 to 0.226], Standard Error of Mean 0.088 — Difference calculated as Tio R5 minus placebo

7. Secondary Outcome: ACQ6 Score Responders
Description: Responder rates based on the ACQ6 score after 12 weeks of treatment. Analysis was performed using the following categories and definitions: responder (change from trial baseline <= -0.5), no change (-0.5 < change from trial baseline <0.5) and worsening (change from trial baseline >= 0.5).
  The ACQ is a scale containing 7 questions, each question has a 7- point scale which ranges from 0 to 6; a score of 0 corresponds to no impairment and a score of 6 corresponds to maximum impairment. ACQ6 is calculated as the mean of the responses to the first 6 questions of the ACQ6.
  No statistical testing was performed on ACQ6 responders.
Time Frame: 12 weeks
Population: Full Analysis Set which included all randomised patients who were dispensed and received at least one documented dose of trial medication.
  Missing data for patients not withdrawn from the study were either categorised as no change or based on available data, withdrawn patients were imputed based upon discontinuation reason.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 135 | 127 | 130
percentage of participants
  Responder | 74.1 | 74.0 | 74.6
  No Change | 23.7 | 19.7 | 23.1
  Worsening | 2.2 | 6.3 | 2.3

8. Secondary Outcome: Control of Asthma as Assessed by ACQ Total Score
Description: Change from baseline in Asthma Control Questionnaire (ACQ) total score measured at week 12.
  The ACQ is a scale containing 7 questions. Each question has a 7 point scale which ranges from 0 to 6. A score of 0 corresponds to no impairment and a score of 6 corresponds to maximum impairment. ACQ total score is calculated as the mean of the responses to all 7 questions.
  The measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 132 | 126 | 130
units on a scale | 1.234 (0.064) | 1.292 (0.066) | 1.270 (0.065)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.4762, Mixed Models Analysis; Mean Difference (Final Values) = 0.058, 95% CI 2-sided [-0.102 to 0.219], Standard Error of Mean 0.082 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.6558, Mixed Models Analysis; Mean Difference (Final Values) = 0.036, 95% CI 2-sided [-0.123 to 0.196], Standard Error of Mean 0.081 — Difference calculated as Tio R5 minus placebo

9. Secondary Outcome: ACQ Total Score Responders
Description: Responder rates based on the ACQ total score after 12 weeks of treatment. Analysis was performed using the following categories and definitions: responder (change from trial baseline ≤-0.5), no change (-0.5 <change from trial baseline <0.5) and worsening (change from trial baseline ≥0.5) No statistical testing was performed for ACQ total score responders.
  The ACQ is a scale containing 7 questions, each question has a 7-point scale which ranges from 0 to 6; a score of 0 corresponds to no impairment and a score of 6 corresponds to maximum impairment.
Time Frame: 12 weeks
Population: Full Analysis Set which included all randomised patients who were dispensed and received at least one documented dose of trial medication. Missing data for patients not withdrawn from the study were either categorised as no change or based on available data. Withdrawn patients were imputed based upon discontinuation reason.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 135 | 127 | 130
percentage of participants
  Responder | 73.3 | 74.8 | 73.1
  No Change | 23.7 | 22.0 | 26.2
  Worsening | 3.0 | 3.1 | 0.8

10. Secondary Outcome: Use of PRN Rescue Medication During the Day
Description: Change from baseline in the number of puffs of rescue medication (salbutamol/albuterol) used during the day (24 hour period) based on the weekly mean at week 12.
  The measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: Full Analysis Set (FAS) was the same as the treated set which included all randomised patients who were dispensed and received at least one documented dose of trial medication. Missing data was imputed by the available data from the patient. Completely missing data were handled by the statistical model.
Measure: Mean (Standard Error); unit: Number of puffs of rescue medication
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 124 | 130
Number of puffs of rescue medication | -0.482 (0.118) | -0.483 (0.122) | -0.540 (0.120)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.9960, Mixed Models Analysis; Mean Difference (Final Values) = -0.001, 95% CI 2-sided [-0.301 to 0.300], Standard Error of Mean 0.153
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.7030, Mixed Models Analysis; Mean Difference (Final Values) = -0.058, 95% CI 2-sided [-0.355 to 0.239], Standard Error of Mean 0.151

11. Secondary Outcome: Use of PRN Rescue Medication During the Daytime
Description: Change from baseline in the number of puffs of rescue medication (salbutamol/albuterol) used during the daytime based on the weekly mean at week 12.
  Measured values presented are actually adjusted means.
Time Frame: Baseline and 12 weeks
Population: as for outcome 10
Measure: Mean (Standard Error); unit: Number of puffs of rescue medication
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 124 | 130
Number of puffs of rescue medication | -0.262 (0.073) | -0.295 (0.075) | -0.312 (0.073)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.7309, Mixed Models Analysis; Mean Difference (Final Values) = -0.032, 95% CI 2-sided [-0.217 to 0.153], Standard Error of Mean 0.094
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.5954, Mixed Models Analysis; Mean Difference (Final Values) = -0.049, 95% CI 2-sided [-0.232 to 0.133], Standard Error of Mean 0.093

12. Secondary Outcome: Use of PRN Rescue Medication During the Night-time
Description: Change from baseline in the number of puffs of rescue medication (salbutamol/albuterol) used during the night-time based on the weekly mean at week 12.
  Measured values presented are actually adjusted means
Time Frame: Baseline and 12 weeks
Population: as for outcome 10
Measure: Mean (Standard Error); unit: Number of puffs of rescue medication
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 124 | 129
Number of puffs of rescue medication | -0.180 (0.064) | -0.092 (0.066) | -0.159 (0.065)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.2841, Mixed Models Analysis; Mean Difference (Final Values) = 0.089, 95% CI 2-sided [-0.074 to 0.252], Standard Error of Mean 0.083
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.7950, Mixed Models Analysis; Mean Difference (Final Values) = 0.021, 95% CI 2-sided [-0.140 to 0.182], Standard Error of Mean 0.082

13. Secondary Outcome: Time to First Severe Asthma Exacerbation During the 12-week Treatment Period.
Description: Time in days to first severe asthma exacerbation during the 12 week treatment period. The median time to first severe asthma exacerbation was not calculable, so the number of patients who experienced a severe asthma exacerbation are presented for the measured values.
  A severe asthma exacerbation was defined as a subgroup of all asthma exacerbations that required an initiation of treatment with systemic corticosteroids for at least 3 days or, in case of ongoing and pre-existing systemic corticosteroid therapy, requiring at least doubling of previous daily doses of systemic corticosteroids for at least 3 days.
Time Frame: 12 weeks
Population: Full Analysis Set (FAS) was the same as the treated set which included all randomised patients who were dispensed and received at least one documented dose of trial medication.
Measure: Number; unit: participants
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 135 | 127 | 130
participants | 1 | 1 | 2
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.9671, Regression, Cox; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.07 to 16.95]
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.5557, Regression, Cox; Hazard Ratio (HR) = 2.06, 95% CI 2-sided [0.19 to 22.70]

14. Secondary Outcome: Analysis of Time to First Asthma Exacerbation During the 12 Week Treatment Period.
Description: Time in days to first asthma exacerbation during the 12 week treatment period. The median time to first asthma exacerbation was not calculable, so the number of patients who experienced an asthma exacerbation are presented for the measured values.
Time Frame: 12 weeks
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 135 | 127 | 130
participants | 25 | 18 | 15
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.3567, Regression, Cox; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.41 to 1.38]
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.1168, Regression, Cox; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.32 to 1.14]

15. Secondary Outcome: Clinically Relevant Abnormalities for Physical Examination, ECG, Vital Signs and Laboratory Tests
Description: Clinically relevant abnormalities for physical examination, ECG, vital signs and laboratory tests. New abnormal findings or worsening of baseline conditions were reported as adverse events.
Time Frame: From first drug administration until 30 days after last drug intake, up to 142 days
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 135 | 127 | 130
percentage of participants
  Peak expiratory flow rate decreased | 9.6 | 7.1 | 3.8
  Blood glucose decreased | 0.0 | 0.8 | 0.0

ADVERSE EVENTS:
Time Frame: From first drug administration until 30 days after last drug intake, up to 142 days
Description: Treated set which included all randomised patients who were dispensed and received at least one documented dose of trial medication.
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Serious Adverse Events (participants affected / at risk) | 0/135 | 1/127 | 2/130
Other Adverse Events (participants affected / at risk) | 23/135 | 23/127 | 16/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Respimat (N=135) | Tio R2.5 (N=127) | Tio R5 (N=130)
Pyoderma (Infections and infestations) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Respimat (N=135) | Tio R2.5 (N=127) | Tio R5 (N=130)
Peak expiratory flow rate decreased (Investigations) | 13 | 9 | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 14 | 14 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BIs intellectual property rights.